CLINICAL TRIAL: NCT01098396
Title: Rasagiline for the Treatment of Gait Disturbances in Patients With Parkinson´S Disease (PD): an Open Label Study
Brief Title: Rasagiline for Gait Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Tanya Gurevich PI, Movement Disorder Unit Dept of Neurology -TASMC
Other Study IDs: TASMC-09-TG-0349
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
Gait disturbances are very common and are a major cause for losing of independency in patients with advanced Parkinson's Disease (PD). The medical treatment of gait disturbances in advanced PD is very difficult and in many cases the classical dopaminergic treatment has no clinical benefit or even can worsen the instability and increase falls. Rasagiline, a new MAO-B inhibitor who has recently been approved all over the world for the treatment of early and late stages PD has been suggested to have a special effect of gait in patients with advanced PD (LARGO sub-study).

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD who experience motor response fluctuations and have gait disturbances at ON and OFF (TUaG >10 secs in ON and 14 secs in OFF) treated with a stable dose of antiparkinsonian medications for the last month. Patients must be able to identify both situations
* Able to walk for 2 minutes at the OFF and ON state
* Non-demented (MMSE= or > to25)

Exclusion Criteria:

* Severe orthopedic problems
* Orthostatic hypotension on basal visit
* Severe, troublesome ON dyskinesias
* Dementia (MMSE <25)
* Major depression
* Active psychosis or on anti-psychotic medications
* Patients who are unlikely to complete the full protocol.
* Patients who have tried rasagiline and stopped because of side effects or lack of symptomatic effect
* Treatment with selegiline for the last 2 months
* Any contraindication according SmPC

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PD
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-05